CLINICAL TRIAL: NCT03884335
Title: Comparison Between Epidural Technique and Mid-axillary Ultrasound-guided TAP Block for Postoperative Analgesia of Laparoscopic Radical Prostatectomy. Impact on Early Discharge
Brief Title: Radical Laparoscopic Prostatectomy. Enhanced Recovery After Surgery (ERAS) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/42
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Prostatectomy
Keywords: Epidural analgesia; Transversus abdominis plane blockade; Laparoscopic prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epidural group (Active Comparator): An epidural catheter was placed at L1-L2 level, and tested, prior to induction. Induction was performed intravenously with fentanyl (1.5mcg•Kg-1), propofol (1.5-2 mg•Kg-1), and rocuronium (0.6 mg•Kg-1). Orotracheal intubation was performed. Prior to skin incision 8 mL of 0.25% levo-bupivacaine were administered epidurally, and a continuous perfusion of 0.125% levo-bupivacaine at 5 mL was started.
  Interventions: Procedure: laparoscopic radical prostatectomy
- TAP group (Experimental): Bilateral Transversus abdominis plane blockade (TAP) was performed following induction of anaesthesia ( the same of epidural group) and prior to skin incision, the high-frequency lineal probe (Sonosite MicroMAXXTM) was placed midway between the costal margin and iliac crest, and transversus abdominis muscle located behind the rectus abdominis and below the IOM. 20 mL of LA (bupivacaine 0.375%) was administered via a 22 gauge Quincke spinal needle inserted in-plane on each side of the abdomen. A successful block was recorded if the plane was seen to expand with fluid under ultrasound vision.
  Interventions: Procedure: laparoscopic radical prostatectomy

INTERVENTIONS:
Procedure: laparoscopic radical prostatectomy — The surgery was carried out by laparoscopy. Intraoperative anesthetic maintenance was performed with TCI of propofol infusion for bispectral index between 40 and 60, restrictive administration of fluids or goal-directed parenteral fluid administration, normothermia, normotension and optimal intraoperative analgesia were maintained following the criteria of ERP. Afterwards, patients were awoken from general anaesthesia and transferred to the post-anaesthesia care unit (PACU) for a 6-hour follow-up prior to transfer to conventional ward.

SUMMARY:
Current trends are based on the implementation of enhanced recovery programs (ERP) for most surgical procedures. The transversus abdominis plane (TAP) block has been demonstrated as an effective analgesic alternative in abdominal surgeries. The goal of this study was to compare analgesic efficacy of the TAP block against epidural technique in patients who underwent laparoscopic radical prostatectomy (LRP) surgery in an ERP setting. This study was performed between October 2016 and May 2018

DETAILED DESCRIPTION:
After approval from Institutional Review Board (approval number 16/42) and compliance with the Declaration of Helsinki; and complying with the information checklist of Consolidated Standards of Reporting trials (CONSORT), informed consent was obtained from all those patients who underwent LRP between October 2016 and May 2018.

Exclusion criteria were: age below 18 years old; American Society of Anaesthesiologists (ASA) score ≥IV; body mass index (BMI) ≥30 Kg/m-2; history of local anaesthetic (LA) allergies; chronic opioid use, coagulopathy; peripheral neuropathy; reconversion to open surgery; or patient's refusal of consent.

Patients were randomized to either TAP or epidural group according to sequential recruitment criteria performed at the pre-operative visit. At this point, age, anaesthesia ASA score and BMI was also recorded.

Management of patients undergoing LRP - intraoperatively All patients underwent combined anaesthesia: either general anaesthesia + epidural; or general anaesthesia + TAP block (TAP group). Patients were premedicated with intravenous midazolam 0.05 mg/Kg-1. In the epidural group, a catheter was placed at L1-L2 level, and tested, prior to induction. Induction was performed intravenously with fentanyl (1.5 mcg/Kg-1), propofol (1.5-2 mg/Kg-1), and rocuronium (0.6 mg/Kg-1). Orotracheal intubation was performed. Prior to skin incision 8 mL of 0.25% levo-bupivacaine were administered epidurally, and a continuous perfusion of 0.125% levo-bupivacaine at 5 mL was started. In the TAP group, a bilateral, ultrasound-guided mid-axillary TAP block was performed immediately after induction (the same as epidural group) but prior to surgery. The high-frequency lineal probe (Sonosite MicroMAXXTM) was placed midway between the costal margin and iliac crest, and transversus abdominis muscle (TAM) located behind the rectus abdominis and below the internal oblique muscle (IOM). 20 mL of LA (bupivacaine 0.375%) was administered via a 22-gauge Quincke spinal needle inserted in-plane on each side of the abdomen. A block was considered successful whenever interfascial local anaesthetic spread was evident under ultrasound vision.

A laparoscopic radical prostatectomy was performed. Intraoperative anaesthetic maintenance was performed with propofol target-controlled infusion (TCI) for bispectral index between 40 and 60. Net zero fluid therapy was maintained, as well as normothermia, normotension and optimal intraoperative analgesia following ERP criteria. After surgery, patients were awoken from general anaesthesia and transferred to the post-anaesthesia care unit (PACU) for a 6-hour follow-up prior to transfer to conventional ward.

The following data was recorded during the intraoperative period: hemodynamic and respiratory parameters, complications related to analgesic technique (vascular puncture, peritoneal or intestinal puncture in the TAP block, number of attempts, impossibility to perform technique), surgery-related complications (bleeding, intestinal, bladder or diaphragmatic perforation), and length of surgery.

Management of patients undergoing LRP - PACU. In the PACU, the patient was kept under observation for 6 hours for pain and bleeding control, as well as hemodynamic and respiratory management. Besides epidural or TAP blockade, standard analgesia was maintained with paracetamol 1g/8h/iv alternate with metamizole 2 g/8h/iv, as well as 2 mg bolus of morphine, if required. If pain was unmanageable, in the epidural group the first option was administration of 8 mL of 0.125% levo-bupivacaine, secondly catheter was re-positioned, and if these options failed, catheter was removed and a morphine infusion was begun. In the TAP group, if rescue morphine bolus (of up to 10mg) was not enough, TAP-block was repeated. If after 20 minutes the patient showed no improvement, morphine infusion was begun. In these cases (both epidural and TAP groups), data was considered as analgesic technique failure.

The following data was recorded during the PACU period: pain as evaluated by the visual analogue scale (VAS) upon rest (VASr) and movement -cough- (VASm) at 1, 2, 3, 4, and 6 hours; mg of morphine administered; failure of analgesic technique (need of morphine PCA); surgical complications; analgesic technique complications (motor blockade, paraesthesias, accidental catheter disconnection); hydric tolerance; postoperative nausea or vomiting (PONV); and time to bowel movement (first flatus after surgery).

Management of patients undergoing LRP - Hospital Ward. After PACU, patients were transferred to conventional hospital ward. During this period, they were followed-up by the hospital's acute pain team, formed by an anaesthesiologist and a specialized nurse.

The following data was registered during this period: VASr and VASm at 12, 18, 24, 36, and 48 hours; time to sitting position and perambulation; PONV; complications of surgical and anaesthetic technique (including infection at this point); mg of morphine administered; failure of analgesic technique (need of morphine PCA); and length of in-hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic radical prostatectomy

Exclusion Criteria:

* anaesthesia ASA score ≥IV;
* body mass index (BMI) ≥30 Kg/m2;
* history of local anaesthesic (LA) allergies, -
* chronic opioid use,
* coagulation alterations (including heparin treatment)
* peripheral neuropathy;
* reconversion to open surgery;
* patient's refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Evolution of postoperative pain over time | Pain was assessed at 1 hour, 2 hours, 3 hours, 4 hours, and 6 hours, and then 12 hours,18 hours, 24 hours, 36 hours and 48 hours
  Pain was evaluated by the visual analogue scale (VAS) upon rest (VASr) and movement -cough- (VASm) at postanesthesia care unit and in the hospital ward. VAS ranges from 0 (no pain) to 10 (maximum pain).

SECONDARY OUTCOMES:
Need for postoperative analgesic medication | up to 6 hours after surgery
  milligrams of morphine administered
Postoperative recovery | up to 24 hours postoperatively
  time to bowel movement (first flatus after surgery)
Evolution till hospital discharge | up to 48 hours postoperatively
  time to sitting position and perambulation